CLINICAL TRIAL: NCT00450294
Title: The Effect of Aortic Infrarenal Clamping and Unclamping On Intraocular Pressure During Abdominal Aortic Aneurysm (AAA) Repair
Brief Title: Intraocular Pressure During Abdominal Aortic Aneurysm (AAA) Repair
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Amit Chopra, Assistant Professor, University of Manitoba
Other Study IDs: B2006:180
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-02

CONDITIONS: Problem With Vision Blindness; Intraocular Pressure; Ischemic Optic Neuropathy
MeSH Terms: conditions — Optic Neuropathy, Ischemic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study will be to answer a clinical question that has not already been investigated; that is, what are the effects of aortic infra-renal clamping and unclamping on intraocular pressure during Abdominal Aortic Aneurysm (AAA) repair? Depending on the results, this study may raise or alleviate concern that vascular surgery for abdominal aortic aneurysm could contribute to early perioperative exacerbation of pre-existing eye disease and increase a patient's vulnerability to developing a type of blindness known as ischemic optic neuropathy. The purpose of this observational study is to evaluate whether intraocular pressure measurements with a handheld tonometer will detect changes in intraocular pressure related to intraoperative events during aortic cross clamping and unclamping that may provide information on causes of perioperative blindness.

DETAILED DESCRIPTION:
Perioperative blindness in nonocular surgery has gained significant clinical interest as an overwhelming complication with an increasing incidence. Initial published studies suggested a rare occurrence with an estimated postoperative visual loss of 0.002% and 0.0008% (1,2). However, retrospective reviews in spinal and cardiac surgery demonstrated higher rates of perioperative blindness; that is, between 0.2% and 0.06% respectively (3,4). The difference in published reports suggests that the true incidence is likely underestimated because of fears regarding litigation, ineffective means of reporting and extra work involved. Fortunately, numerous case reports and series in the middle to late 1990s were published; prompting the American Society of Anesthesiologists (ASA) Committee on Professional Liability to establish the ASA Postoperative Visual Loss Registry (POVL) in 1999 as a medium to collect confidential, comprehensive perioperative data on patients developing postoperative blindness.

The POVL registry, along with other case series, has demonstrated that the most common cause of visual loss is non-arteritic ischemic optic neuropathy (5,6,7). Perioperative non-arteritic ischemic optic neuropathy (ION) is a consequence of patient and surgery specific factors that results from hypoperfusion and infarction of the optic nerve head (8). Anatomical factors such as variation in the number of short posterior ciliary arteries (sPCA) supplying the optic nerve head, location of sPCA watershed zone, and small optic cup to disk ratio increase susceptibility to optic nerve ischemia (8,9). Surgery specific factors involve profound blood loss, anemia, hypotension, prone positioning and duration of surgery (5,6,7,10). The interaction of these surgical variables and patient specific anatomical factors can decrease ocular perfusion pressure (the difference between mean arterial pressure and intraocular pressure) and result in ION (11).

Based on the determinants of ocular perfusion pressure (OPP), low mean arterial pressure (MAP) and/or high intraocular pressure (IOP) can decrease OPP and lead to ION. Therefore, it is necessary to investigate changes in IOP incurred from different types of surgery that may increase vulnerability to developing ION. Normal IOP is between 12 - 20 mm Hg. Studies have been published assessing intraocular changes with prone positioning, laparoscopic surgery and cardiopulmonary bypass (12,13,14). However, there has been no literature evaluating intraocular pressure during abdominal aortic aneurysm (AAA) repair. AAA repair is a high-risk surgery associated with blood loss, hypotension and has been reported in a case series associated with ION (6). The surgery involves clamping and unclamping of the aorta to facilitate excision of the aneurysm and graft repair. Aortic cross clamping and unclamping is an intense physiologic insult affecting venous return, systemic vascular resistance, cardiac output, and acid base status. These physiologic changes are further pronounced with more proximal cross-clamping and longer duration. Because infrarenal abdominal aortic aneurysms are the most common type of AAA repair, we will be assessing IOP with patients undergoing elective infrarenal abdominal aortic reconstruction.

Infrarenal aortic cross clamping is associated with increases in venous return, central venous pressure and arterial blood pressure (15). The hemodynamic changes with infrarenal unclamping entail decreases in venous return, central venous pressure and arterial blood pressure (15). The determinants of intraocular pressure involve extraocular muscle tone, aqueous flow, choroidal blood volume and central venous pressure (16). The volume redistribution proximal to the aortic cross-clamp should cause a rise in venous pressure, increase resistance to aqueous drainage and increase choroidal blood volume thereby increasing intraocular pressure. However, after aortic unclamping, choroidal blood volume and IOP should decrease as venous return and central venous pressure decline. Therefore, our hypothesis is that IOP will be increased during aortic cross clamping and decreased following aortic unclamping.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to St. Boniface General Hospital for elective AAA repair requiring an arterial line, central line and general anesthesia will be eligible for inclusion in this study.

Exclusion Criteria:

* . The exclusion criteria for this study are:

  1. Patients with a history of acute or chronic eye disease
  2. Allergy to topical ophthalmologic anesthesia
  3. Patients receiving nitrous oxide, ketamine or succinylcholine during anesthesia
  4. If the surgical procedure will require the aorta to be re-clamped following unclamping, those patients will also be excluded
  5. Patients that are VRE+ or MRSA+ will be excluded for infection control purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with known infrarenal abdominal aortic aneurysm for open repair will be screened through the preadmission anesthetic clinic. If they do not meet exclusion criteria and have signed informed consent for the the study, they will be enrolled to assess for changes in intraocular pressure during open abdominal aortic aneurysm repair.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-03; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Chopra, M.D., Principal Investigator — University of Manitoba, Department Of Anesthesiology, Faculty of Medicine
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Roth S, Thisted RA, Erickson JP, Black S, Schreider BD. Eye injuries after nonocular surgery. A study of 60,965 anesthetics from 1988 to 1992. Anesthesiology. 1996 Nov;85(5):1020-7. doi: 10.1097/00000542-199611000-00009. PMID 8916818
- [Background] Warner ME, Warner MA, Garrity JA, MacKenzie RA, Warner DO. The frequency of perioperative vision loss. Anesth Analg. 2001 Dec;93(6):1417-21, table of contents. doi: 10.1097/00000539-200112000-00013. PMID 11726416
- [Background] Stevens WR, Glazer PA, Kelley SD, Lietman TM, Bradford DS. Ophthalmic complications after spinal surgery. Spine (Phila Pa 1976). 1997 Jun 15;22(12):1319-24. doi: 10.1097/00007632-199706150-00008. PMID 9201834
- [Background] Nuttall GA, Garrity JA, Dearani JA, Abel MD, Schroeder DR, Mullany CJ. Risk factors for ischemic optic neuropathy after cardiopulmonary bypass: a matched case/control study. Anesth Analg. 2001 Dec;93(6):1410-6, table of contents. doi: 10.1097/00000539-200112000-00012. PMID 11726415
- [Background] Lee LA, Roth S, Posner KL, Cheney FW, Caplan RA, Newman NJ, Domino KB. The American Society of Anesthesiologists Postoperative Visual Loss Registry: analysis of 93 spine surgery cases with postoperative visual loss. Anesthesiology. 2006 Oct;105(4):652-9; quiz 867-8. doi: 10.1097/00000542-200610000-00007. PMID 17006060
- [Background] Brown RH, Schauble JF, Miller NR. Anemia and hypotension as contributors to perioperative loss of vision. Anesthesiology. 1994 Jan;80(1):222-6. doi: 10.1097/00000542-199401000-00033. No abstract available. PMID 8291715
- [Background] Myers MA, Hamilton SR, Bogosian AJ, Smith CH, Wagner TA. Visual loss as a complication of spine surgery. A review of 37 cases. Spine (Phila Pa 1976). 1997 Jun 15;22(12):1325-9. doi: 10.1097/00007632-199706150-00009. PMID 9201835
- [Background] Hayreh SS, Jonas JB. Optic disc morphology after arteritic anterior ischemic optic neuropathy. Ophthalmology. 2001 Sep;108(9):1586-94. doi: 10.1016/s0161-6420(01)00649-2. PMID 11535455
- [Background] Beck RW, Servais GE, Hayreh SS. Anterior ischemic optic neuropathy. IX. Cup-to-disc ratio and its role in pathogenesis. Ophthalmology. 1987 Nov;94(11):1503-8. PMID 3684223
- [Background] Williams EL, Hart WM Jr, Tempelhoff R. Postoperative ischemic optic neuropathy. Anesth Analg. 1995 May;80(5):1018-29. doi: 10.1097/00000539-199505000-00029. No abstract available. PMID 7726399
- [Background] Hayreh SS. Anterior ischemic optic neuropathy. Clin Neurosci. 1997;4(5):251-63. PMID 9292252
- [Background] Cheng MA, Todorov A, Tempelhoff R, McHugh T, Crowder CM, Lauryssen C. The effect of prone positioning on intraocular pressure in anesthetized patients. Anesthesiology. 2001 Dec;95(6):1351-5. doi: 10.1097/00000542-200112000-00012. PMID 11748391
- [Background] 13 Kayacan N, Gulbin A, Akar M, Karsli B. The effect of pneumoperitoneum and head-down position on intraocular pressure. Gynaecological Endoscopy 2002;11:383-87.
- [Background] Larkin DF, Connolly P, Magner JB, Wood AE, Eustace P. Intraocular pressure during cardiopulmonary bypass. Br J Ophthalmol. 1987 Mar;71(3):177-80. doi: 10.1136/bjo.71.3.177. PMID 3828271
- [Background] Gelman S. The pathophysiology of aortic cross-clamping and unclamping. Anesthesiology. 1995 Apr;82(4):1026-60. doi: 10.1097/00000542-199504000-00027. No abstract available. PMID 7717537
- [Background] Murphy DF. Anesthesia and intraocular pressure. Anesth Analg. 1985 May;64(5):520-30. No abstract available. PMID 3158256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten patients were recruited into the study after informed consent at the preoperative anesthetic clinic during a twelve month period.
Pre-assignment Details: Because this is a purely OBSERVATIONAL STUDY, there was no group assignment. All patients enrolled in the study were assigned to one group, that is, all patients had intraocular pressure measurements performed.
Groups:
- Longitudinal Study Group: This study is an OBSERVATIONAL STUDY. Ten patients were enrolled to determine what happens to eye pressure during surgery for abdominal aortic aneurysm repair. Therefore, all ten patients had intraocular pressure measurements made at different event intervals to determine if there was a change in intraocular pressure compared to their baseline intraocular pressure that was taken before surgery. No active intervention was performed to the patients based on intraocular pressure as clinicians were blinded to the intraocular pressure values.Measurement of Central venous pressure at event intervals during abdominal aortic aneurysm repair. Data are presented as mean +/- standard error.
Period: Overall Study
Arm/Group | Longitudinal Study Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Longitudinal Group: This study is an observational longitudinal design. Ten patients were enrolled to determine what happens to eye pressure during surgery for abdominal aortic aneurysm repair. Therefore, all ten patients had intraocular pressure measurements made at different event intervals to determine if there was a change in intraocular pressure compared to their baseline intraocular pressure that was taken before surgery. No active intervention was performed to the patients based on intraocular pressure as clinicians were blinded to the intraocular pressure values.
Arm/Group | Longitudinal Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  Canada | 10
Cross Clamp Duration [Mean (Standard Deviation); unit: min] | 58 (15.3)
Preop Right Intraocular Pressure [Mean (Standard Deviation); unit: mm Hg] | 16.9 (2.6)
Preop Left Intraocular Pressure [Mean (Standard Deviation); unit: mm HG] | 16.7 (2.7)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 27.3 (3.4)
Abdominal Aortic Aneurysm Size [Mean (Standard Deviation); unit: cm] | 5.7 (0.5)
Cerebrovascular Accident (CVA) [Number; unit: participants]
  HAS CVA | 4
  No CVA | 6
Diabetes mellitus [Number; unit: participants]
  HAS DM | 10
  NO DM | 0
Hypertension [Number; unit: participants]
  HAS HTN | 10
  NO HTN | 0
Hyperlipidemia [Number; unit: participants]
  HAS Hyperlipidemia | 10
  NO Hyperlipidemia | 0
Epidural [Number; unit: participants]
  Epidural | 10
  NO Epidural | 0
Cumulative Crystalloid [Mean (Standard Deviation); unit: L] | 2.84 (0.13)
Vasopressor infusion [Number; unit: participants]
  Vasopressor Infusion | 10
  NO vasopressor infusion | 0
Mannitol [Number; unit: participants]
  Received Mannitol | 10
  N) Mannitol | 0
ASA Physical Status [Number; unit: participants] — ASA physical status classification is a score given to the patient by the anesthesiologist following a preoperative assessment. It pertains to the patient's preoperative fitness. The full categorization scheme is as follows:
  1. Healthy person.
  2. Mild systemic disease.
  3. Severe systemic disease.
  4. Severe systemic disease that is a constant threat to life.
  5. A moribund person who is not expected to survive without the operation.
  participants
    ASA I (healthy person) | 0
    ASA II (mild systemic disease) | 0
    AASA III (Severe systemic disease) | 10
    ASA IV (Severe systemic disease, constant threat) | 0
    ASA V (moribund person) | 0

OUTCOME MEASURES:

1. Primary Outcome: Right Intraocular Pressure During Various Event Intervals in Open Abdominal Aortic Aneurysm Surgery.
Description: Intraocular pressure measurements were made with a tonometer. These measurements were recorded and kept blinded from the clinicians.
Time Frame: Measurements made at baseline, post induction preincision, 1 min post clamp, 5 min post clamp, 1 min pre unclamp, 1 min post unclamp, 5 min post unclamp, skin closure
Population: The analysis was per protocol.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Longitudinal Group: This study is an OBSERVATIONAL STUDY. Ten patients were enrolled to determine what happens to eye pressure during surgery for abdominal aortic aneurysm repair. Therefore, all ten patients had intraocular pressure measurements made at different event intervals to determine if there was a change in intraocular pressure compared to their baseline intraocular pressure that was taken before surgery. No active intervention was performed to the patients based on intraocular pressure as clinicians were blinded to the intraocular pressure values.
Arm/Group | Longitudinal Group
Number analyzed (Participants) | 10
mm Hg
  Preoperative | 16.9 (0.75)
  Pre-induction | 13.8 (0.75)
  1 min post clamp | 14.6 (0.75)
  5 min post clamp | 13.5 (0.75)
  1 min before unclamp | 14.1 (0.75)
  1 min following unclamp | 14.4 (0.75)
  5 min following unclamp | 15 (0.75)
  Skin closure | 14.1 (0.75)
Statistical Analysis 1: Comparison: Longitudinal Group; Repeated measures anova with post hoc t-tests using tukey's correction; Test type: Superiority or Other; p < 0.001, ANOVA — That the means at the different timepoints would not all be equal

2. Primary Outcome: Left Intraocular Pressure
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Longitudinal Study Group: This study is an observational longitudinal design. Ten patients were enrolled to determine what happens to eye pressure during surgery for abdominal aortic aneurysm repair.
Arm/Group | Longitudinal Study Group
Number analyzed (Participants) | 10
mm Hg
  Preoperative | 16.7 (0.57)
  Pre-incision | 15 (0.57)
  1 min post clamp | 14.7 (0.57)
  5 min post clamp | 13.7 (0.57)
  1 min before unclamp | 14.6 (0.57)
  1 min following unclamp | 15.1 (0.57)
  5 min following unclamp | 15.3 (0.57)
  Skin closure | 14.7 (0.57)
Statistical Analysis 1: Comparison: Longitudinal Study Group; Repeated measures anova with post hoc t-tests using tukey's correction; Test type: Superiority or Other; p < 0.001, ANOVA — That the means at the different timepoints would not all be equal

ADVERSE EVENTS:
Arm/Group | Longitudinal Group
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
There were no limitations to trial during course of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No